CLINICAL TRIAL: NCT04835337
Title: Investigating the Health Benefits of Indoor Air Filtration Among Children: a Randomized Crossover Trial in Jiaozuo, China
Brief Title: The Health Benefits of Indoor Air Filtration Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tiantian Li (Other Government)
Responsible Party: Sponsor-Investigator, Tiantian Li, professor, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 202032
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Protective Effect of Air Purifier on Children's Health
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air purifier (Experimental): Participants in this group receive an intervention of real air purifiers placed in the indoor environment.
  Interventions: Behavioral: Air Purifiers
- Control (Sham Comparator): Participants in this group receive an intervention of sham air purifiers, we just remove the filter in the purifiers, and the other treatments are the same as the real purification group.
  Interventions: Behavioral: Sham Air Purifiers

INTERVENTIONS:
Behavioral: Air Purifiers — Students are divided into two groups: intervention group and control group. The intervention team places an air purifier in the indoor environment to intervene. All the indoor environment of the group use the same qualified air purifier, and all participants and research staffs are blinded to the group assignment.
  Arms: Air purifier
Behavioral: Sham Air Purifiers — The control group is also intervened. The intervention is to place a sham air purifier (remove the filter screen) in the indoor environment, and all the indoor environment use the same air purifier as the intervention group. All participants and research staffs are blinded to the group assignment.
  Arms: Control

SUMMARY:
This study aims to explore the health benefits of air purifier on the impact of air pollutants on children's health.

DETAILED DESCRIPTION:
From April 2021 to December 2021, researchers conduct a randomized double-blind crossover trial on about 100 healthy children in Jiaozuo City, Henan Province. The children are divided into two groups according to their classes and alternated the use of true or sham purifiers devices, including air purifiers and fresh air ventilation. Air purifiers are installed in the classroom and bedrooms of the children. Fresh air ventilation is installed in the classroom. A total of 4 epidemiological surveys are conducted on the subjects, with an interval of 60 days or more. All participants and research staffs were blinded to the group assignment. In addition, air pollutant exposure monitoring, questionnaire surveys, physical examinations, and biological sample collection are conducted on the research subjects each time. The biological samples are further tested for the concentration levels of related biomarkers such as the respiratory system, cardiovascular system, metabolic system, and nervous system. Furthermore, comprehensive evaluation of children's behavioral ability is also carried out. Ambient PM2.5 and indoor PM2.5 exposure concentrations are monitored in the study.

ELIGIBILITY:
Inclusion Criteria:

* 10 ≤ 12 years old
* Volunteer to participate in this study

Exclusion Criteria:

* Current and past medical history, including asthma, childhood diabetes, childhood hypertension, behavior-related diseases
* Students who plan to transfer or move within six months
* Unable to cooperate with follow-up

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Changes of FEV1 | Baseline and at the end of each 60 days intervention period
  The forced expiratory volume in 1 s (FEV1) is measured using a smart spirometer (Model A1, BreathHome, China) supervised by professional medical staff. Before the pulmonary function test, subjects will practice several times by themselves. During the examination, each subject stands and clamps the nose clip, and repeats the test, with the best result as the criterion. FEV1 reflect pulmonary function.
Changes of FVC | Baseline and at the end of each 60 days intervention period
  The forced vital capacity (FVC) is measured using spirometer (Model A1, BreathHome, China). FVC reflects the expiratory resistance of large airways.
Changes of FEV1/FVC ratio | Baseline and at the end of each 60 days intervention period
  The FEV1/FVC ratio is measured using smart spirometer (Model A1, BreathHome, China). FEV1/FVC ratio reflects the status of airway obstruction.
Changes of PEF | Baseline and at the end of each 60 days intervention period
  The peak expiratory flow (PEF) is measured using smart spirometer (Model A1, BreathHome, China). PEF reflects airway patency and respiratory muscle strength.
Changes of FEF25-75% | Baseline and at the end of each 60 days intervention period
  The forced expiratory flow at 25-75% of FVC (FEF25-75%) is measured using smart spirometer (Model A1, BreathHome, China). FEF25-75% reflects the small airway obstruction.
Changes of MEF75% | Baseline and at the end of each 60 days intervention period
  The maximal expiratory flow at 75% of FVC (MEF75%) is measured using smart spirometer (Model A1, BreathHome, China). MEF75% reflects the terminal stage of expiratory flow rate.
Changes of MEF50% | Baseline and at the end of each 60 days intervention period
  The maximal expiratory flow at 50% of FVC (MEF50%) is measured using smart spirometer (Model A1, BreathHome, China). MEF50% reflects the interim stage of expiratory flow rate.
Changes of MEF25% | Baseline and at the end of each 60 days intervention period
  The maximal expiratory flow at 25% of FVC (MEF25%) is measured using smart spirometer (Model A1, BreathHome, China). MEF25% reflects the early stage of expiratory flow rate.
Changes of FeNO | Baseline and at the end of each 60 days intervention period
  Use NIOX VERO Sensor to measure fractional exhaled nitric oxide (FeNO) as a biomarker for airway inflammation level. After deep breathing, the subjects gently inhaled into the device. The instrument showed FeNO level of the subjects.
Changes of FeCO | Baseline and at the end of each 60 days intervention period
  Use Pico Smokerlyzer to measure fractional exhaled carbon monoxide (FeCO). After deep breathing, the subjects held their breath for 15 seconds and then gently inhaled into the device. The instrument showed FeCO level and the estimated value of carboxyhemoglobin in blood.
Changes of Blood Pressure | Baseline and at the end of each 60 days intervention period
  The professional staffs wrap the BP cuff around the left upper arm of children to measure BP using the Omron electronic sphygmomanometers (OMROM, J751). BP is measured at 2-minute intervals, with a total of three measurements taken. If the difference of BP values between the last two measurements exceeds 5 mmHg, additional measurements are performed. Each child is allowed to measure BP at least three times and up to five times. The BP indicators includes SBP, DBP, MAP and PP.
Changes of heart rate variability | Baseline and at the end of each 60 days intervention period
  The trained staffs conduct a 3-minute comprehensive assessment using the handheld electrocardiographic recorder-CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measured HRV. The time-domain indicators include standard deviation of all normal-to-normal intervals (SDNN), the root mean square of successive differences between adjacent normal cycles (rMSSD), the percentage of adjacent NN interval differences greater than 50 ms (pNN50); and the frequency-domain indicators include very low frequency (VLF), low frequency (LF), high frequency (HF), the ratio of LF to HF (LF/HF). To eliminate possible error, subjects are conducted by the same trained staff using the same instrument.
Changes of PR interval | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the interval of the beginning of the P wave to the beginning of the QRS complex (PR interval).
Changes of QRS duration | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the interval of the beginning of Q wave to the end of the S wave (QRS duration).
Changes of QT interval | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the interval from the onset of the QRS complex to the end of the T wave (QT interval).
Changes of QTc interval | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the QT correction for rate (QTc interval).
Changes of RV5 | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the amplitude of the R-wave in lead V5 (RV5).
Changes of SV1 | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the S-wave depth in lead V1 (SV1).
Changes of RV5+SV1 | Baseline and at the end of each 60 days intervention period
  The trained staff use a 12-lead electrocardiogram (ECG) monitor to measure the participants' the sum of the R-wave amplitude in lead V5 and the S-wave amplitude in lead V1(RV5+SV1).
Changes of academic performance | Baseline and at the end of each 60 days intervention period
  The assessment of academic performance consists of standardised scores (maths, chinese and total) and the relative rank of the scores within grade. Standardised scores are converted from raw scores (with minimum value of 0 and maximum of 100) according to the number of exams and classes, indicating the position of the sample value in the normal distribution curve, with higher value showing better outcome. Rankings are converted from place rankings of raw values, with lower value showing better outcome.

SECONDARY OUTCOMES:
Changes of CRP | Baseline and at the end of each 60 days intervention period
  Detect the concentration of C-reactive protein in blood sample to examine the different level of inflammation between the group of intervention and control.
Changes of 8-OHdG | Baseline and at the end of each 60 days intervention period
  Detect the concentration of 8-hydroxydeoxyguanosine (8-OHdG) in urine sample as a marker of generalized, cellular oxidative stress to DNA.
Changes of metabolites in exhaled breath condensate | Baseline and at the end of each 60 days intervention period
  Collect the exhaled breath condensate and identify the metabolites of exhaled breath condensate using Ultra-high performance liquid chromatography-tandem mass spectrometry.
Changes of the role of alertness | Baseline and at the end of each 60 days intervention period
  Alertness can be measured by the Attention Network Test and reflects an individual's acquisition and maintenance of a state of alertness to a particular type of information or target.
Changes of the role of orientation | Baseline and at the end of each 60 days intervention period
  Orientation can be measured by the Attention Network Test and reflects an individual's selective attention to externally useful information.
Changes of the role of conflict | Baseline and at the end of each 60 days intervention period
  Conflict can be measured by the Attention Network Test and reflects an individual's ability to process conflicting information.
Changes of Wisconsin Card Sorting Test indicators | Baseline and at the end of each 60 days intervention period
  WCST contains absolute indicators of cognitive executive functioning which include level of conceptualisation, persistence and set maintenance. The cognitive absolute indicators include conceptual thinking includes complete correct (TC), complete error (TE), non-persistent error (NPE), conceptual level response (CLR) and category completed (CC), persistence includes persistent response (PR) and persistent error (PE), and pooling maintenance includes inability to maintain pooling (FM).WCST percentage metrics are similar in meaning to the absolute metrics, and can be categorised into the level of conceptualisation and the Two dimensions of persistence. Cognitive percentage indicators include conceptual thinking consists of total correct percentage (%TC), total error percentage (%TE), non-persistent error percentage (%NPE), and conceptual level response percentage (%NPE); persistence consists of persistent response percentage (%PR) and persistent error percentage (%PE).
Changes of the position total number | Baseline and at the end of each 60 days intervention period
  The position total number is the number of all position-related stimuli during the N-back test. The subjects need to remember how each position changed and judge whether a duplicate position stimulus appeared after N rounds.
Changes of the position number correct | Baseline and at the end of each 60 days intervention period
  The position number correct is the number of times during the N-back test that the subjects were able to correctly judge whether or not a repeated position appeared in N rounds. A higher number correct indicates that the tester performed better in remembering and recognising the location.
Changes of the position percentage correct | Baseline and at the end of each 60 days intervention period
  Changes of position percentage correct is the accuracy of the -N-back test subjects in position-related tasks, expressed as a percentage. It is calculated as (number of locations correct ÷ total number of location stimuli) × 100%. A high rate of correctness indicates that the subjects' accuracy in location memory is high.
Changes of the color total number | Baseline and at the end of each 60 days intervention period
  The color total number is the number of all colour-related stimuli during the -N-back test. The subjects were required to remember the colour changes and determine whether a repeated colour stimulus has occurred after N-backs.
Changes of the color number correct | Baseline and at the end of each 60 days intervention period
  The color number correct is the number of times during the N-back test that the subjects were able to correctly judge whether a repeated colour appeared or not in N rounds. A higher correct count indicates that the tester performed better in colour memory and recognition.
Changes of the color percentage correct | Baseline and at the end of each 60 days intervention period
  Changes of color percentage correct is is the subjects' accuracy in colour-related tasks during the N-back test, expressed as a percentage. It is calculated as (number of colours correct ÷ total number of colour stimuli) × 100%. A high rate of correctness indicates that the subjects' accuracy in colour memory is high.
Changes of the shape total number | Baseline and at the end of each 60 days intervention period
  The shape total number is the number of all shape stimuli during the N-back test. The subjects need to remember the shape changes and judge whether a repeated shape stimulus has appeared after the N-back.
Changes of the shape number correct | Baseline and at the end of each 60 days intervention period
  The shape number correct is the number of times during the N-back test that the subjects were able to correctly judge whether or not a repeated shape appeared in N rounds. A higher number correct indicates that the subjects performed better in shape memory and recognition.
Changes of the shape percentage correct | Baseline and at the end of each 60 days intervention period
  Changes of shape percentage correct is the subjects' accuracy in shape-related tasks during the N-back test, expressed as a percentage. It is calculated as (number of shapes correct ÷ total number of shape stimuli) × 100%. A high rate of correctness indicates that the subjects' accuracy in shape memory is high.
Changes of proteins in serum | Baseline and at the end of each 60 days intervention period
  Collect peripheral venous blood, extract the serum, and identify the proteins of serum samples using 4D-label free technology.
Changes in biomarkers identified from other omics | Through study completion, up to 10 years
  Collect peripheral venous blood, exhaled breath condensate, urine, saliva, oral cells, oral swabs, nasal swabs, skin swabs, nails and feces samples, then identify the biomarkers by conducting transcriptomic, microbiome analyses, etc.
Changes in other targeted biomarkers of interest | Through study completion, up to 10 years
  Collect peripheral venous blood, exhaled breath condensate, urine, saliva, oral cells, oral swabs, nasal swabs, skin swabs, nails and feces samples, then identify the other targeted biomarkers of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Tiantian Li, Study Director — National Institute of Environmental Health, Chinese Center for Disease Control and Prevention
Locations (1):
- National Institute of Environmental Health, Chinese Center for Disease Control and Prevention, Beijing, China

REFERENCES:
- [Derived] Lei J, Sun Q, Chen R, Zhu Y, Zhou L, Xue X, Fang J, Du Y, Wang Y, Li T, Kan H. Respiratory Benefits of Multisetting Air Purification in Children: A Cluster Randomized Crossover Trial. JAMA Pediatr. 2025 Feb 1;179(2):122-128. doi: 10.1001/jamapediatrics.2024.5049. PMID 39621320

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04835337/Prot_SAP_003.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT04835337/ICF_001.pdf